CLINICAL TRIAL: NCT06744751
Title: A Randomsized Controlled Study on the Effects of Combined Fecal Microbiota Transplantation on Gut Microbiota and Eating Disorder Symptoms in Patients With Anorexia Nervosa
Brief Title: A Study on the Effects of Combined FMT on Gut Microbiota and Eating Disorder Symptoms in AN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-28
Record Dates: First submitted 2024-11-07; First posted 2024-12-20 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia nervosa; Tretment of Anorexia nervosa; Gastrointestinal symptoms in Anorexia nervosa; Gut microbiota
MeSH Terms: conditions — Anorexia Nervosa | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fecal Microbiota Transplantation (Active Comparator): The FMT capsules used in this study contain processed, frozen stool from healthy donors, providing gut microbiota from these individuals. The FMT capsules meet relevant manufacturing standards. Patients take the capsules twice daily, with a dose of 6 or 10 capsules per day, over a period of 6 days (for a total of 72 or 120 capsules). Select the capsule dosage based on age. For children under 18 years old, take 10 capsules at a time. For adults aged 18 and above, take 6 capsules at a time.
  Interventions: Biological: Fecal Microbiota Transplantation
- Placebo (Placebo Comparator): The placebo capsules, manufactured by the same company, are identical in appearance, size, color, dosage form, weight, and taste to the FMT capsules. Starch is used as the main ingredient to mimic the FMT capsules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation — Patients take the capsules twice daily, with a dose of 6 or 10 capsules per day, for a total of 6 days (72 or 120 capsules in total). Select the capsule dosage based on age. For children under 18 years old, take 10 capsules at a time. For adults aged 18 and above, take 6 capsules at a time. Both the FMT and placebo capsules are identical in appearance, size, color, form, weight, and taste, with the placebo containing starch as the main ingredient.
  Arms: Fecal Microbiota Transplantation
Drug: Placebo — Manufactured by the same company, the placebo capsules contain starch as the main ingredient and are identical in appearance, size, color, dosage form, weight, and taste to the FMT capsules. They are administered twice daily, 6 or 10 capsules per dose (selected by age), for 6 days.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to determine if Fecal Microbiota Transplantation (FMT) is effective in treating Anorexia Nervosa (AN). The study will also explore how FMT works. The main questions it aims to answer are:

1. What is the efficacy of combined FMT treatment in patients with AN?
2. What is the relationship between treatment efficacy and changes in gut microbiota, and what mechanisms underlie the effects of FMT in treating AN? Researchers will compare FMT to a placebo (a look-alike substance that contains no active ingredients) to see if FMT is effective in treating AN.

Participants will:

* Be hospitalized
* Take FMT or placebo daily for 6 days
* Provide stool and blood samples before and after FMT
* Visit the clinic every 4 weeks for check-ups and tests

DETAILED DESCRIPTION:
Anorexia Nervosa (AN) is a chronic, challenging psychiatric disorder characterized by an intense fear of gaining weight, extreme weight loss, severe malnutrition, and physical wasting. The core behavioral trait of AN is a "persistent restriction of energy intake," which results in low body weight, malnutrition, and, in severe cases, death due to multiple organ failure. Consequently, AN is considered the most fatal mental disorder. With globalization and rapid economic development in China, dieting and weight loss have become fashionable. A domestic survey found that 49.9% to 55.7% of female college students engage in dieting and weight loss behaviors, and the prevalence of AN in China has been increasing rapidly. Thus, AN is becoming a significant public health issue in China.

More than 90% of AN patients experience functional gastrointestinal symptoms (FGS), including bloating, constipation, and difficulty swallowing. These FGS are largely associated with disordered eating behaviors. For example, patients with restrictive eating often prefer high-fiber, low-fat, and low-carbohydrate foods, which can lead to symptoms such as early satiety, constipation, and flatulence. Therefore, disordered eating behavior can contribute to abnormal gastrointestinal function, while, conversely, disordered GI function can exacerbate the severity of AN, hinder patients from resuming normal eating habits, and impact the effectiveness of clinical treatment. Recent studies increasingly suggest that gut microbes play an essential role in influencing GI symptoms in psychiatric disorders.

The human gastrointestinal tract hosts billions of microorganisms, with a total gene count about 150 times greater than that of the human genome. These microorganisms are closely linked to the regulation of gastrointestinal function and have also been shown to influence mood, eating behavior, appetite, and nutrient metabolism. Researchers have discovered that Nod2 receptors expressed by inhibitory neurons in the hypothalamus and arcuate nucleus can directly sense cytosolic peptides produced by bacteria, regulating feeding behavior and suggesting that gut microbes may influence appetite through the brain-gut axis. Cross-sectional studies have found abnormalities in gut flora composition or metabolites in AN patients, while longitudinal studies have shown that the abundance of gut flora increases after weight regain in AN patients; however, flora diversity and gastrointestinal symptoms do not fully return to normal. This suggests that, while body weight may normalize, the gut microbiome remains "unhealthy."

Fecal Microbiota Transplantation (FMT) involves transplanting healthy intestinal flora into a patient's gut. FMT primarily treats digestive diseases like intestinal infections, irritable bowel syndrome, Crohn's disease, and chronic diarrhea, effectively relieving symptoms such as constipation and diarrhea. FMT has also been used to treat neuropsychiatric disorders like autism, mood disorders, ADHD, and sleep disorders. Studies have shown that FMT can alleviate symptoms of depression, anxiety, and sleep disturbances caused by chronic stress, reduce inflammatory responses to slow the progression of Alzheimer's disease, and improve symptoms in patients with autism spectrum disorder (ASD). Although some case reports describe FMT's application in AN patients, there is still a lack of extensive randomized controlled trials to validate its efficacy.

Currently, no studies have explored the role of FMT combined with conventional treatments in improving AN's clinical symptoms. Given that mood and GI symptoms are common comorbidities of AN, and there is no effective pharmacologic treatment for these symptoms, FMT offers a promising new strategy to enhance clinical outcomes as a supportive treatment for AN.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 12-35 years, meets DSM-5 diagnostic criteria for anorexia nervosa.
* BMI > 14 kg/m²; for children/adolescents, BMI > the 0.3 percentile for their age.
* Presence of digestive symptoms (e.g., constipation, bloating, diarrhea).
* Duration of the disease (since the onset of dieting and weight loss) is less than two years.
* Each patient must understand the nature of this study and sign an informed consent form.

Exclusion Criteria:

* Co-morbid severe mental disorders such as schizophrenia, bipolar disorder, intellectual disability, persistent delusional disorder, schizoaffective disorder, or organic mental disorders.
* Substance abusers/addicts, individuals with a high suicide risk, or those with strong destructive impulses or antisocial behavior.
* Those with severe low body mass anorexia nervosa (e.g., blood pressure < 80/50 mmHg, heart rate < 40 beats/min, weight loss > 1 kg per week, or those requiring assistance in sitting or squatting in a prone position).
* Patients with severe somatic diseases or comorbidities, including:
* Organic intestinal lesions such as congenital megacolon, intestinal obstruction, or intussusception.
* Previous pathological intestinal inflammatory conditions such as inflammatory bowel disease.
* History of traumatic brain injury, cerebral palsy, encephalitis, or other organic brain disorders.
* Severe hepatic or renal insufficiency (defined as levels greater than three times the upper limit of normal).
* Pregnant or breastfeeding women.
* Use of medications such as probiotics or antibiotics that clearly affect the intestinal flora within 1 months prior to the visit or during the treatment.
* Any other reason that the investigator deems unsuitable for participation in this clinical trial.

Ages: 12 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Hight | baseline，follow-up (4,8,12 week)
  Measurement of morning height will be taken using the same height-measuring device.
Weight | baseline，follow-up (4,8,12 week)
  Morning fasting weight will be measured using the same scale.

SECONDARY OUTCOMES:
Eating Disorder Examination Questionnaire 6.0(EDEQ-6.0) | baseline，follow-up (4,8,12 week)
  The Eating Disorder Examination Questionnaire 6.0 (EDE-Q 6.0) is a self-assessment questionnaire based on the Eating Disorder Examination (EDE). It evaluates the primary behavioral and psychological characteristics of eating disorders, measuring both the frequency and intensity of symptoms to assess disorder severity. The questionnaire includes four subscales: dietary restriction, eating concerns, body image concerns, and weight concerns.
Gastrointestinal Symptom Rating Scale(GSRS) | recuitment， follow-up（4、8、12 week）
  The Gastrointestinal Symptom Rating Scale (GSRS) consists of 15 items designed to assess a patient's gastrointestinal symptoms over the past week. Each question is scored based on the degree, frequency, duration, mitigating factors, and impact on social activities, using a scale from 0 to 3, where 0 indicates no symptoms and 3 indicates very severe symptoms. The scores for each question are summed to give a total score, with a minimum of 0 and a maximum of 45. Higher scores indicate more severe gastrointestinal symptoms.
Hamilton Depression Scale (HAMD) | baseline，follow-up（4、8、12 week）
  The Hamilton Depression Scale (HAMD) is an external evaluation scale used to assess a patient's depression symptoms. The scale consists of 24 items. Most of the questions are scored on a 0-4 point scale, while questions 4, 5, 6, 12, 13, 14, 16, 17, 18, and 21 are scored on a 0-2 point scale (a three-level scoring system). The total score ranges from a minimum of 0 to a maximum of 76, with higher scores indicating more severe depression symptoms.
Patient Health Questionnaire-9 (PHQ-9) | baseline, follow-up(4, 8, 12 week)
  The Patient Health Questionnaire-9 (PHQ-9), based on the DSM-IV diagnostic criteria, consists of 9 items, using a four-point rating scale of 0 to 3. Scores ranging from 5 to 9 indicate mild depression, 10 to 14 indicate moderate depression, 15 to 19 indicate moderately severe depression, and 20 to 27 indicate severe depression.
Clinical Global Impression (CGI) | baseline, follow-up(4, 8, 12 week)
  This scale is divided into three items: severity of the disease, overall efficacy assessment, and efficacy index. The severity of illness uses an 8-point rating scale from 0 to 7, with 0 indicating no disease and 7 indicating extremely severe. The global improvement assessment uses an 8-point rating scale from 0 to 7, with 0 indicating no assessment and 7 indicating severe deterioration. The efficacy index uses a four-level rating, with efficacy divided into four levels: 4 indicates marked improvement, with symptoms completely or largely disappearing; 1 indicates no change or deterioration; side effects are rated into four levels: 4 indicates serious or even life-threatening side effects occurred; 1 indicates no side effects.
Fecal microbiota | baseline，follow-up（4、12week）
  Change in diversity and composition of the fecal microbiota as assessed by macrogenomic sequencing of feces.
Short-chain fatty acids | baseline，follow-up（4、12 week）
  Blood was collected and centrifuged to obtain serum, which was then tested for short-chain fatty acids.

IPD SHARING:
Plan to Share IPD: No